CLINICAL TRIAL: NCT03985085
Title: PrEP, Sexually Transmitted Infections, Contraception, Hepatitis B Virus, and Sexual Health for Female Sex Workers in Côte d'Ivoire
Brief Title: Sexual and Reproductive Health (Including PrEP and HBV) for Female Sex Workers in Côte d'Ivoire
Acronym: ANRS 12381
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Programme PAC-CI (Unknown); Aprosam, San Pedro (Unknown); Institut de Recherche pour le Developpement (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ANRS 12381 PRINCESSE
Record Dates: First submitted 2019-03-13; First posted 2019-06-13 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: HIV Infections; Viral Hepatitis B; Sexually Transmitted Diseases; Contraception
Keywords: female sex workers
MeSH Terms: conditions — HIV Infections; Hepatitis B; Sexually Transmitted Diseases | interventions — Reproductive Health Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental)
  Interventions: Other: Comprehensive package of sexual and reproductive health services

INTERVENTIONS:
Other: Comprehensive package of sexual and reproductive health services — Implementation of a comprehensive sexual and reproductive health care package for female sex workers in Côte d'Ivoire, combining an HIV PrEP offer (for HIV- FSW) with early treatment of HIV+ FSW, management of HBV infection (testing, vaccination and treatment), testing and treatment of sexually transmitted infections (STIs) and their consequences, a contraception offer, a quarterly screening of pregnancies, menstrual management counselling and identification of addiction.
  This healthcare package will be available both in mobile clinics organized for a quarterly follow-up (10 intervention sites, each site being visited every two weeks) and in the fixed clinic of the partner community-based NGO, at the discretion of each female participant.

SUMMARY:
The PRINCESSE study will implement a comprehensive package of services in sexual and reproductive health for female sex workers in the region of San Pedro in Cote d'Ivoire, including screening, prevention and treatment for HIV, viral hepatitis B, sexually transmitted infections and family planning. All services will be available in mobiles clinics operating on prostitution sites and organized for a chronic follow-up of participants.

DETAILED DESCRIPTION:
PRINCESSE is a single-arm interventional cohort of 500 female sex workers (FSWs) in San Pedro, Cote d'Ivoire (400 HIV-negative FSW and 100 HIV-positive FSW).

It consists in the implementation of a comprehensive sexual and reproductive health care package for female sex workers in Côte d'Ivoire, combining an HIV PrEP offer (for HIV- FSW) with early treatment of HIV+ FSW, management of HBV infection (testing, vaccination and treatment), testing and treatment of sexually transmitted infections (STIs) and their consequences, a contraception offer, a quarterly screening of pregnancies, menstrual management counselling and identification of addiction.

This healthcare package will be available both in mobile clinics organized for a quarterly follow-up (10 intervention sites, each site being visited every two weeks) and in the fixed clinic of the partner community-based NGO, at the discretion of each female participant.

The main objective is to develop, document and analyze a community-based healthcare package combining testing, prevention tools including pre-exposure prophylaxis (PrEP), immediate HIV treatment, management of Hepatitis B virus and sexual and reproductive health (SRH)

Specific objectives are:

1. To analyse access to care and retention into care, and more generally female participants' healthcare trajectories through a quarterly follow-up of FSWs (infected with HIV or not)
2. To measure female participants' health outcome over time of clinical, behavioural and social indicators
3. To assess PrEP initiation, use and adherence
4. To compare HIV management in the PRINCESSE system with the existing routine treatment and care
5. To measure HBV testing, vaccination and treatment, as part of a decentralised management integrated with HIV PrEP, and possible interactions between HIV PrEP and HBV infection
6. To document the unexpected consequences (positive or negative) of PRINCESSE system on the everyday life of female participants in particular, and on the sex industry in general
7. To evaluate the impact of vaginal microbiota on bacterial sexually transmitted infections, human papillomavirus (HPV) infections and associated cervical lesions; the impact of the HPV type distribution on the vaccinal strategy and the added value of HPV PCR for the primary screening of cervical cancer; and the impact of antimicrobial resistance on the STI guidelines.
8. Assess the a priori acceptability and appropriateness of different forms of long-acting PrEP for different sex workers profiles.

Four data collection devices are included in the cohort: (i) clinical and safety data, (ii) socio-behavioural questionnaires, (iii) biological data, and (iv) in-depth interviews with female participants.

Eight additional data collections are scheduled outside the cohort itself: (i) capture of medical and activity records of Aprosam for PRINCESSE participants; (ii) capture of medical records of HIV+ FSW patients not participating in the PRINCESSE cohort and routinely examined by the NGO partner; (iii) in-depth interviews with key informants in the FSW community; (iv) in-depth interviews with PRINCESSE follow-up actors (peer educators and caregivers) (v) individual biographical interviews with female sex workers recruited by Aprosam and Espace Confiance about long-acting PrEP, supplemented by (vi) focus group discussions with female sex workers; (vii) focus group discussions with sex workers assigned men at birth; (viii) individual interviews with community actors.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman over 18 years of age
* Self-reporting as being a sex worker
* Wishing to enrol in a regular clinical follow-up
* Agreeing to participate in the study and signing the informed consent form
* Regardless of HIV status (infected or not)
* Whether or not the participant has already taken antiretrovirals
* Whether or not the participant is already followed by Aprosam

Exclusion Criteria:

* Participation in another biomedical and/or behavioural study on HIV, viral hepatitis or Sexually Transmitted Infections

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-11-26 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Completion rate of quarterly visits | up to 24 months
  Proportion of completed study visits
Proportion with at least one diagnosed STI | up to 24 months
Occurrence of an unwanted pregnancy in the last 12 months | up to 24 months
Initiation of PrEP | over 24 months
  Among those eligible for PrEP, proportion having initiating PrEP
Adherence to PrEP | up to 24 months
  among those on PrEP, proportion being adherent (measured through self-report, pill count and drug detection in plasma)
Number of participants in HIV care at 18 months (retention) | 18 months
  Among those HIV-infected at baseline
Occurrence of virological failure | over 24 months (survival analysis)
  Among those HIV-infected and having initiated antiretroviral treatment, proportion with two consecutive detectable viral loads
HBV vaccination rate | over 24 months
  among those needing hepatitis B vaccination, proportion with complete vaccination (3 doses if HIV-negative, 8 doses if HIV-positive) at the end of the trial
Initiation and number of participants on TDF (retention) for patients with a treatment for HBV mono-infection | over 24 months
  among those with positive HBs-antigen and a F3-F4 fibrosis
Proportion with increase in transaminase level (flares) after PrEP discontinuation | within 12 months after PrEP discontinuation
  Among those who started and stopped PrEP and with a positive HBs antigen
Number of adverse social events occurring in the daily life of participants | over 24 months
  Assessment of adverse social events occurring in the daily life of participants
Composition of the vaginal microbiota | up to 12 months
  Percentage of cervical lesions at M0 and M12
Percentage of HPV infection and distribution of subtypes | up to 12 months
Percentage of resistant bacterial STIs | up to 12 months
  Percentage of M.genitalium infections with mutations resistant to macrolide and fluoroquinolone at M0 and M12 Percentage of N.gonorrhoeae infections with resistance genes resistant to fluoroquinolone, ceftriaxone and cyclin at M0 and M12
Percentage of acceptability of different forms of long-acting PrEP for different sex workers profiles | over 12 months
  Percentage of acceptability will be measured with in-depth individual interviews conducted with sex workers using a semi-structured interview guide including a biographical grid

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Larmarange, PhD, Principal Investigator — Institut de Recherche pour le Développement (IRD); Sege Eholié, MD PhD, Principal Investigator — Programme PAC-CI
Locations (1):
- Aprosam, San-Pédro, Côte d’Ivoire

IPD SHARING:
Plan to Share IPD: Yes
The detailed IPD will be developed in the first year of project implementation to determine exact data that will be shared.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: within 24 months after trial's end

REFERENCES:
- [Derived] Becquet V, Nouaman M, Plazy M, Agoua A, Zebago C, Dao H, Montoyo A, Jary A, Coffie PA, Eholie S, Larmarange J; the ANRS 12381 PRINCESSE team. A community-based healthcare package combining testing and prevention tools, including pre-exposure prophylaxis (PrEP), immediate HIV treatment, management of hepatitis B virus, and sexual and reproductive health (SRH), targeting female sex workers (FSWs) in Cote d'Ivoire: the ANRS 12381 PRINCESSE project. BMC Public Health. 2021 Dec 4;21(1):2214. doi: 10.1186/s12889-021-12235-0. PMID 34863122